CLINICAL TRIAL: NCT06888739
Title: Development and Validation of Interpretable Machine Learning Models Incorporating Paraspinal Muscle Quality for to Predict Cage Subsidence Risk Followingposterior Lumbar Interbody Fusion
Status: Completed | Type: Observational
Sponsor: Hao Liu (Other)
Responsible Party: Sponsor-Investigator, Hao Liu, Department of Orthopedics, The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu Province, China, First Affiliated Hospital of Suzhou Medical College
Organization: First Affiliated Hospital of Suzhou Medical College (Other)
Other Study IDs: （2025）Lun Yan Grant No. 220; （2025）Lun Yan Grant No. 220 (Other: Ethics Committee of the First Affiliated Hospital of Soochow University)
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Lumbar Diseases; Cage; Machine Learning
Keywords: Degenerative lumbar disease; Cage subsidence; Machine learning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The study does not include biological samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Subsidence Group: Group A (n = 390): Lost IH value <2 mm.Cage subsidence was defined as a lost IH value ≥2 mm during the follow-up period
  Interventions: Procedure: MR4
- Subsidence Group: Lost IH value ≥2 mm.Cage subsidence was defined as a lost IH value ≥2 mm during the follow-up period
  Interventions: Procedure: MR4

INTERVENTIONS:
Procedure: MR4 — The study is a clinical retrospective study and does not involve any interventional measures.

SUMMARY:
The study focuses on identifying risk factors for cage subsidence after posterior lumbar interbody fusion (PLIF) and developing an interpretable machine learning model to predict these risks. It analyzes patients from two large teaching hospitals, using clinical, radiographic, and surgical parameters, including paraspinal muscle indices and bone density markers. A web-based application was developed to facilitate real-time clinical risk assessments using the machine learning model, enhancing surgical planning and reducing subsidence risks.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed lumbar disc herniation, spinal stenosis, or spondylolisthesis based on clinical and imaging findings;
2. patients who failed conservative treatment for ≥3 months or experienced recurrence and underwent surgery for the first time;
3. minimum 12-month follow-up.

Exclusion Criteria:

1. prior spinal surgery;
2. spinal deformity or severe instability;
3. lumbar tuberculosis, infection, tumor, or severe bone destruction;
4. incomplete or lost follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included patients with degenerative lumbar diseases who underwent single-level PLIF at the First and Second Affiliated Hospitals of Soochow University (January 2018-October 2023).A total of 620 patients from the First Affiliated Hospital comprised the training set, while 100 patients from the Second Affiliated Hospital formed the external validation set. The study adhered to the Declaration of Helsinki and was approved by the institutional ethics committee.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Bone density imaging indicator: Vertebral Bone Quality (VBQ) | Preoperative measurement for PLIF (Posterior Lumbar Interbody Fusion)
  VBQ is calculated by dividing the mean T1 signal intensity (L1-L4) by the cerebrospinal fluid (CSF) signal at L3

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University Medical Record and Imaging System, Jiangsu, SuZhou, China

IPD SHARING:
Plan to Share IPD: Yes
Before January 1,2026;in the form of paper. The original data of the trial will be uploaded to Genome Sequence Archive (GSA) (ngdc.cncb.ac.cn)